CLINICAL TRIAL: NCT06219538
Title: DAISY Uterine Drain: Device Evaluation With Standard Wall Suction
Brief Title: DAISY Uterine Drain Device Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Raydiant Oximetry, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CP2400
Record Dates: First submitted 2024-01-03; First posted 2024-01-23 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Cesarean Section Complications; Post Partum Hemorrhage; Uterine Atony With Hemorrhage; Uterine Bleeding
Keywords: uterine drain; PPH
MeSH Terms: conditions — Postpartum Hemorrhage; Uterine Hemorrhage

STUDY DESIGN:
Intervention Model Description: The participants consist of women undergoing planned CD for reasons unrelated to this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Interventional (Experimental): Ten women in whom the Daisy Drain is placed.
  Interventions: Device: DAISY Uterine Drain

INTERVENTIONS:
Device: DAISY Uterine Drain — Insertion of the DAISY Uterine Drain and connection to wall suction in women who have undergone a Caesarean Delivery,

SUMMARY:
The goal of this study is to obtain user feedback while placing and observing the DAISY uterine drain with wall suction. This study defines the obstetrical surgeons as "users" and the patients in whom the drain is placed as "participants." Participants are pregnant women who are undergoing cesarean delivery (CD), who have not entered active labor, who have consented to drain placement and who have met all the inclusion/exclusion criteria. Users are staff or fellow obstetrical surgeons who will use the drain and provide the evaluation.

DETAILED DESCRIPTION:
Postpartum hemorrhage (PPH) is the leading cause of maternal mortality worldwide. (D'Alton 2020). It is estimated that 14 million cases of PPH occur each year worldwide (Rath, 2011). In the United States, PPH causes up to 12% of maternal deaths and is the leading cause of death occurring on the day of delivery (ACOG 2017; Butwick 2019; Evensen 2020; Hawkins 2020). According to the American College of Obstetricians and Gynecologists (ACOG), between 54% and 93% of PPH-associated mortality may be preventable while 70-80% of PPH is due to abnormal uterine tone (atony) (ACOG 2017). Atony involves a deficient response to physiological signals that promote uterine contraction and blood vessel compression after delivery. Contraction of the myometrium compresses the blood vessels supplying the placental bed and thereby causes mechanical hemostasis. Uterine atony following CD is a relatively common problem in the non-laboring patient because contraction of the myometrium is almost entirely absent. Restoring uterine tone can be addressed through 1) medication, 2) surgery, or 3) mechanical means. Post-partum unrecognized uterine hemorrhage due to a closed or narrow cervix that allows blood to collect in a patient undergoing a CD could lead to complications such as dangerously low blood pressure. The DAISY drain is intended to provide a channel through the cervix for fluid drainage after pelvic surgery. The DAISY device consists of a soft silicone drainage tube (proximal end) attached to a semi-flexible catheter, inserted through the hysterotomy created at the time of the CD. The DAISY drain is placed intraoperatively after delivery of the placenta, stabilization of the patient, and cleansing of the uterine cavity but prior to closure of the hysterotomy. The drain is placed through the hysterotomy and threaded through the cervix and vaginal canal, out the introitus, so the distal end is accessible outside of the body. In this study, the drain is placed on continuous suction according to the IFU for the first two postoperative hours or more if required. At the end of the 2-hour period, the uterus is evaluated by manual palpation and abdominal ultrasound. The abdominal ultrasound is performed to document device placement and to assess uterine involution, approximate uterine size and uterine cavity size, presence of intrauterine clots or retained products of conception. The trained user removes the drain after at least two hours post-surgery based on clinical management. Suction is discontinued before removal. One method of determining if the drain is no longer needed is by checking and documenting uterine tone. If uterine tone has returned to normal as assessed by palpation, the DAISY drain may be removed.

ELIGIBILITY:
Inclusion Criteria:

* The participants consist of women undergoing planned CD for reasons unrelated to this study.

Exclusion Criteria:

* Known intrauterine or cervical pathology that would interfere with device placement and/or use
* Ongoing intrauterine pregnancy
* Untreated uterine rupture
* Unresolved uterine inversion
* Current cervical cancer
* Current purulent infection of vagina, cervix, or uterus
* Retained products of conception
* Arterial bleeding requiring surgical or angiographic embolization
* Indication for hysterectomy
* Lack of study consent or unable to provide informed consent,
* Any condition (temporary or permanent) in which the investigator or user deems the patient unsuitable for the study procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only adult women over the age of eighteen can be included.
Enrollment: 10 (Actual)
Dates: Start 2024-05-22 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
Device evaluation | Immediately post procedure
  This is a prospective, single-arm, device evaluation study of device use by five (5) obstetrical surgeons placing the drain with low-level suction in up to ten (10) women undergoing elective, non-emergent cesarean delivery. A user questionnaire is filled out. The questionnaire asks users to evaluate various aspects of the device. The DAISY drain and Instructions for Use (IFU) are evaluated qualitatively for the following including:
  * ease of drain placement by obstetrician-surgeon
  * appropriate size of drain
  * appropriate final location of the deployed drain and incidence of improper placement
  * ease of drain connection to suction tubing
  * ease of drain removal
  * perceived effectiveness of suction
  * clarity of the IFU

CONTACTS AND LOCATIONS:
Overall Officials: Tetsuya Kawakita, MD, Principal Investigator — Eastern Virginia Medical School
Locations (1):
- Eastern Virginia Medical School, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kawakita T, Ray N, Brennan M, Rosen M, Saade G. A Uterine Suction Device to Prevent Postpartum Hemorrhage in Scheduled Cesarean Delivery: A Pilot Study. Am J Perinatol. 2025 Dec 4. doi: 10.1055/a-2752-8798. Online ahead of print. PMID 41285413